CLINICAL TRIAL: NCT01004198
Title: A Multi-center, Randomized, Double-blind, Controlled Dose-finding Study to Evaluate the Safety and Efficacy of MP4OX Treatment Plus Standard of Care in Severely Injured Trauma Patients With Lactic Acidosis Due to Hemorrhagic Shock
Brief Title: Phase IIa Study of MP4OX in Traumatic Hemorrhagic Shock Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sangart (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRA-204
Record Dates: First submitted 2009-10-28; First posted 2009-10-29 (Estimated); Last update posted 2013-08-19 (Estimated); Status verified 2013-08

CONDITIONS: Shock, Hemorrhagic; Shock, Traumatic; Acidosis, Lactic
Keywords: Trauma; Hemorrhage; Hemorrhagic shock; Lactic acidosis; Oxygen carriers; Oxygen therapeutics; Hemoglobin solutions; Hemoglobin substitutes; Red cell substitutes; PEG-hemoglobin
MeSH Terms: conditions — Shock, Hemorrhagic; Shock, Traumatic; Acidosis, Lactic; Wounds and Injuries; Hemorrhage | interventions — maleimide-polyethylene glycol-modified hemoglobin, MP4; PEG-hemoglobin; Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- MP4OX - 250 (Experimental): 250 mL dose
  Interventions: Drug: MP4OX
- MP4OX - 500 (Experimental): 500 mL dose
  Interventions: Drug: MP4OX
- Ringers Lactate solution (Active Comparator): 500 mL dose
  Interventions: Drug: Ringers Lactate solution

INTERVENTIONS:
Drug: MP4OX — 4.3 g/dL PEG-Hb solution in lactated electrolyte solution
  Other Names: MP4; MalPEG-Hb; PEG-Hb; Pegylated-Hb
  Arms: MP4OX - 250
Drug: MP4OX — 4.3 g/dL PEG-Hb solution in lactated electrolyte solution
  Other Names: MP4; MalPEG-Hb; PEG-Hb; Pegylated-Hb
  Arms: MP4OX - 500
Drug: Ringers Lactate solution — Ringers Lactate solution for Injection
  Other Names: Lactated Ringers; Hartmann's solution
  Arms: Ringers Lactate solution

SUMMARY:
MP4OX is a novel oxygen therapeutic agent specifically developed to perfuse and oxygenate tissue at risk for ischemia and hypoxia. MP4OX is a pegylated hemoglobin-based colloid and and as a result of its molecular size and unique oxygen dissociation characteristics, targets oxygen delivery to ischemic tissues by selectively off-loading oxygen in tissues predisposed to low oxygen tension. Sangart is currently evaluating MP4OX to reduce organ dysfunction and failure in trauma patients with lactic acidosis due to severe hemorrhagic shock.

DETAILED DESCRIPTION:
Acute traumatic injury, including both blunt and penetrating injury, is often associated with severe bleeding which can lead to hemorrhagic shock. During shock, inadequate perfusion of critical organs can lead to local ischemia and tissue hypoxia (insufficient oxygenation), which can be detected by an increase in serum lactate levels. Despite optimal care, more than 10% of trauma victims who reach hospital alive will die, and many will suffer from organ failure. Death and significant, persistent morbidity are consequences of trauma, and traumatic injuries are associated with lost productivity, reduced quality of life, and direct costs to patients and health care systems worldwide. Current therapies, which also include blood transfusion, are aimed at supporting failing organs, but a therapeutic agent that could help to quickly restore adequate oxygenation may be beneficial to prevent or shorten duration of organ failure and improve patient outcome.

Direct support for the proposed clinical application to use MP4OX in resuscitation from hemorrhage is found in preclinical animal studies. Using a pig model of uncontrolled hemorrhage and resuscitation, survival was greater and restoration of hemodynamics and acid-base status were improved with MP4OX relative to an equivalent volume of crystalloid, pentastarch, or unmodified hemoglobin. Administration of MP4OX improved 24-hour survival, stabilized cardiac output and arterial pressure at nearly normal levels, and reduced lactate levels more effectively than the control fluids. Importantly, these benefits of MP4OX were observed with or without co-administration of autologous blood, suggesting that blood alone was not sufficient to achieve complete resuscitation, and that the effects of MP4OX appear to be additional to those of blood.

ELIGIBILITY:
Inclusion Criteria:

* Adult male or female (surgically sterile or post-menopausal or confirmed not to be pregnant)
* Trauma injury (blunt and/or penetrating) resulting in lactic acidosis due to hemorrhagic shock (blood lactate level ≥ 5 mmol/L; equivalent to ≥ 45 mg/dL)
* Informed consent obtained before any study-related activities

Exclusion Criteria:

* Not expected to survive 24 hours after randomization
* Evidence of severe traumatic brain injury as defined by any one of the following: Known non-survivable head injury or open brain injury; Glasgow Coma Score (GCS) = 3, 4 or 5, or known AIS = 5 if GCS > 5; Immediate open intracranial operation; Abnormal physical exam indicative of severe CNS or spinal injury
* Significant ongoing uncontrolled hemorrhage where control of bleeding is not expected within 2 hours of randomization
* Cardiac arrest prior to dosing
* Estimated time from injury to dosing > 4 hours
* Estimated time from hospital admission to randomization > 2 hours
* Known or suspected pregnancy (confirmed by urine test)
* Previous participation in this study
* Professional or ancillary personnel involved with this study
* Receipt of any investigational drug(s) within 30 days prior to study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Serum lactate clearance | 2 hours

SECONDARY OUTCOMES:
All-cause mortality | 28 days
Ventilator-free days | 28 days
ICU-free days | 28 days
Hospital-free days | 28 days
Sepsis-related Organ Failure Assessment (SOFA) score | Daily
Modified Denver score | Daily
Composite endpoint of Time to Complete Organ Failure Resolution (CTCOFR) | At 14 and 21 days

CONTACTS AND LOCATIONS:
Overall Officials: Karim Brohi, MD, Principal Investigator — The Royal London Hospital
Locations (13):
- France (4):
  - Centre Hospitalier de Bicêtre, Le Kremlin-Bicêtre
  - CHRU de Lille - Hôpital Claude Huriez, Lille
  - Hôpital Dupuytren, Limoges
  - Hôpital Pitié-Salpêtrière, Paris
- Germany (2):
  - Charité Campus Virchow Klinikum, Berlin
  - Klinikum der Johann-Wolfgang-Goethe-Universität, Frankfurt
- South Africa (6):
  - Netcare Union Hospital, Alberton
  - Charlotte Maxeke Johannesburg Hospital, Johannesburg
  - Netcare Milpark Hospital, Johannesburg
  - Netcare Unitas Hospital, Centurian, Pretoria
  - Steve Biko Academic Hospital, Pretoria
  - Chris Hani Baragwanath Hospital, Soweto
- The Royal London Hospital, London, United Kingdom

REFERENCES:
- [Background] Olofsson C, Ahl T, Johansson T, Larsson S, Nellgard P, Ponzer S, Fagrell B, Przybelski R, Keipert P, Winslow N, Winslow RM. A multicenter clinical study of the safety and activity of maleimide-polyethylene glycol-modified Hemoglobin (Hemospan) in patients undergoing major orthopedic surgery. Anesthesiology. 2006 Dec;105(6):1153-63. doi: 10.1097/00000542-200612000-00015. PMID 17122578
- [Background] Olofsson C, Nygards EB, Ponzer S, Fagrell B, Przybelski R, Keipert PE, Winslow N, Winslow RM. A randomized, single-blind, increasing dose safety trial of an oxygen-carrying plasma expander (Hemospan) administered to orthopaedic surgery patients with spinal anaesthesia. Transfus Med. 2008 Feb;18(1):28-39. doi: 10.1111/j.1365-3148.2007.00811.x. PMID 18279190
- [Background] Young MA, Lohman J, Malavalli A, Vandegriff KD, Winslow RM. Hemospan improves outcome in a model of perioperative hemodilution and blood loss in the rat: comparison with hydroxyethyl starch. J Cardiothorac Vasc Anesth. 2009 Jun;23(3):339-47. doi: 10.1053/j.jvca.2008.08.006. Epub 2008 Oct 22. PMID 18948027
- [Background] Young MA, Riddez L, Kjellstrom BT, Winslow RM. Effect of maleimide-polyethylene glycol hemoglobin (MP4) on hemodynamics and acid-base status after uncontrolled hemorrhage in anesthetized swine: comparison with crystalloid and blood. J Trauma. 2007 Dec;63(6):1234-44. doi: 10.1097/TA.0b013e31815bd7b0. PMID 18212644
- [Background] Young MA, Riddez L, Kjellstrom BT, Bursell J, Winslow F, Lohman J, Winslow RM. MalPEG-hemoglobin (MP4) improves hemodynamics, acid-base status, and survival after uncontrolled hemorrhage in anesthetized swine. Crit Care Med. 2005 Aug;33(8):1794-804. doi: 10.1097/01.ccm.0000172648.55309.13. PMID 16096458
- [Background] Drobin D, Kjellstrom BT, Malm E, Malavalli A, Lohman J, Vandegriff KD, Young MA, Winslow RM. Hemodynamic response and oxygen transport in pigs resuscitated with maleimide-polyethylene glycol-modified hemoglobin (MP4). J Appl Physiol (1985). 2004 May;96(5):1843-53. doi: 10.1152/japplphysiol.00530.2003. Epub 2004 Jan 16. PMID 14729723
- [Background] Vandegriff KD, Winslow RM. Hemospan: design principles for a new class of oxygen therapeutic. Artif Organs. 2009 Feb;33(2):133-8. doi: 10.1111/j.1525-1594.2008.00697.x. PMID 19178457
- [Background] Vandegriff KD, Malavalli A, Mkrtchyan GM, Spann SN, Baker DA, Winslow RM. Sites of modification of hemospan, a poly(ethylene glycol)-modified human hemoglobin for use as an oxygen therapeutic. Bioconjug Chem. 2008 Nov 19;19(11):2163-70. doi: 10.1021/bc8002666. PMID 18837531
- [Background] Tsai AG, Cabrales P, Manjula BN, Acharya SA, Winslow RM, Intaglietta M. Dissociation of local nitric oxide concentration and vasoconstriction in the presence of cell-free hemoglobin oxygen carriers. Blood. 2006 Nov 15;108(10):3603-10. doi: 10.1182/blood-2006-02-005272. Epub 2006 Jul 20. PMID 16857991
- [Background] van der Linden P, Gazdzik TS, Jahoda D, Heylen RJ, Skowronski JC, Pellar D, Kofranek I, Gorecki AZ, Fagrell B, Keipert PE, Hardiman YJ, Levy H; 6090 Study Investigators. A double-blind, randomized, multicenter study of MP4OX for treatment of perioperative hypotension in patients undergoing primary hip arthroplasty under spinal anesthesia. Anesth Analg. 2011 Apr;112(4):759-73. doi: 10.1213/ANE.0b013e31820c7b5f. Epub 2011 Feb 11. PMID 21317165
- See also: www.Sangart.com — http://www.sangart.com